CLINICAL TRIAL: NCT07285265
Title: A Randomized, Blinded and Positive-Control Phase I Clinical Trial to Evaluate the Immunogenicity and Safety of Lyophilized Herpes Zoster mRNA Vaccine in Adults Aged 40 Years or Above
Brief Title: Phase I Clinical Trial of Lyophilized Herpes Zoster mRNA Vaccine in Adults Aged 40 Years or Above
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Suzhou Abogen Biosciences Co., Ltd. (Industry)
Collaborators: Abogen Biosciences (Shanghai) Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: ABO1108-101
Record Dates: First submitted 2025-12-03; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Varicella-zoster Virus
MeSH Terms: conditions — Chickenpox

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort 1: Dose level A in adults aged 40 years or above (Other): Two injections of Dose level A of ABO1108 or placebo or active competitor given approximately 60 days apart
  Interventions: Biological: ABO1108; Drug: Placebo; Biological: SHINGRIX
- Cohort 2: Dose level B in adults aged 40 years or above (Other): Two injections of Dose level B of ABO1108 or placebo or active competitor given approximately 60 days apart
  Interventions: Biological: ABO1108; Drug: Placebo; Biological: SHINGRIX
- Cohort 3: Dose level C in adults aged 40 years or above (Other): Two injections of Dose level C of ABO1108 or placebo or active competitor given approximately 60 days apart
  Interventions: Biological: ABO1108; Drug: Placebo; Biological: SHINGRIX

INTERVENTIONS:
Biological: ABO1108 — Formulation for injection
Drug: Placebo — 0.9% sodium chloride (normal saline) injection
Biological: SHINGRIX — • Formulation for injection

SUMMARY:
The primary objective of this study is to evaluate the tolerability, reactogenicity and safety of 2 injections (approximately 2 months apart) of three different dose levels of ABO1108 in adults aged 40 years or above.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign the Informed Consent Form (ICF) approved by the Ethics Committee and agree to participate in the trial before undergoing any trial procedures.
2. Healthy adults ≥40 years of age, participants with underlying diseases that are stably controlled may be accepted.
3. Willing to and physically able to communicate with the investigators, understand and comply with protocol required follow-up, simple self-observation and recording using the Diary Card.
4. Male participants (and their female partners) and female participants of childbearing potential agree to continue effective contraception through 12 months following vaccination.

Exclusion Criteria:

1. Acute illness or fever on the day of vaccination or within 3 days prior to vaccination, or use of anti-inflammatory, anti-allergy, antibiotic, or antiviral medications due to physical discomfort.
2. Clinically significant abnormal vital signs, including but not limited to:

   * Resting pulse rate <50 beats per minute or >100 beats per minute
   * Systolic blood pressure ≥140 mmHg or diastolic blood pressure ≥90 mmHg for participants aged 40-59, or systolic blood pressure ≥150 mmHg or diastolic blood pressure ≥90 mmHg for participants aged ≥60
   * Body mass index (BMI) ≤18 kg/m² or ≥30 kg/m²
3. Clinically significant abnormalities of laboratory indicators or 12-lead ECG during the screening period.
4. Female participants known to be pregnant or breastfeeding, or positive pregnancy test for women of childbearing potential.
5. History of allergy to the investigational product or its excipients, or severe allergic reactions to other vaccines, foods, or medications.
6. History of herpes zoster at any previous time, history of varicella or close contact with varicella/herpes zoster patients within the past year.
7. Previous vaccination with herpes zoster or varicella vaccine (including marketed or investigational vaccines) or planned vaccination during the trial period.
8. Use or planned use of any vaccine other than the investigational products through 30 days prior to and 30 days after vaccinations in this trial.
9. Current participation in another clinical trial within 6 months prior to vaccination or planned participation before the end of this trial.
10. Clinician-diagnosed coagulation abnormalities.
11. Known medical history or diagnosis confirming the subject has a condition affecting immune system function.
12. History of myocarditis, pericarditis, or idiopathic cardiomyopathy, or presence of any condition that may increase the risk of myocarditis or pericarditis.
13. Severe or uncontrolled respiratory, cardiovascular, neurological, hematological, lymphatic, hepatic, renal, metabolic, or skeletal diseases; known severe congenital malformations; developmental disorders; or clinically diagnosed severe chronic conditions that may affect trial outcomes.
14. Current infectious period of any communicable disease, acute infection, or acute phase of chronic infection, or ongoing anti-tuberculosis treatment; or prior positive test for hepatitis B surface antigen, hepatitis C virus antibody, or Treponema pallidum antibody.
15. Past or current diagnosis of neurological or psychiatric disorders, or family history of neurological/psychiatric disorders; or other neurological conditions deemed unsuitable for trial participation by the investigator.
16. Long-term use of immunosuppressants or immunomodulators through 6 months prior to and one month after the last vaccination, excluding topical medications. Topical medications should not exceed recommended doses or induce systemic exposure.
17. Treatment with immunoglobulins and/or blood products or blood donation through 3 months prior to and 3 months after the last vaccination in this trial.
18. Suspected or known alcohol dependence or drug abuse, which may affect safety assessment or trial compliance.
19. Planned long-term or permanent relocation away from the trial site area before trial completion.
20. Investigators, sponsors, and contract research organization (CRO) staff directly involved in the trial.

Other circumstances deemed unsuitable for trial participation by the investigator.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2025-05-27 (Actual); Primary Completion 2025-11-06 (Actual); Study Completion 2026-10-15 (Estimated)

PRIMARY OUTCOMES:
Incidence of solicited AEs and ARs after each dose | up to day 74 (14 days after each dose)
Incidence of unsolicited AEs and ARs after each dose | up to day 90 (30 days after each dose)

CONTACTS AND LOCATIONS:
Locations (1):
- Rongshui Miao Autonomous County Center for Disease Control and Prevention, Liuchow, Rongshui, China

IPD SHARING:
Plan to Share IPD: No